CLINICAL TRIAL: NCT06504186
Title: A Prospective, Single-arm Clinical Study of the Use of Blinatumomab in Patients With NGS-MRD Relapsed B-ALL After Autologous/Allogeneic Transplantation
Brief Title: The Use of Blinatumomab in Patients With NGS-MRD Relapsed B-ALL After Autologous/Allogeneic Transplantation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IIT2024044
Record Dates: First submitted 2024-07-10; First posted 2024-07-16 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-06

CONDITIONS: B-ALL
MeSH Terms: interventions — blinatumomab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NGS-MRD relapsed B-ALL after autologous/allogeneic transplantation (Other): * Ph-negative B-ALL: bephedolumab (≥ 45 kg: 9 mcg/d D1-2, 28 mcg/d D3-14 or 28 mcg/d D1-14; < 45 kg: 5 mg/m2/d D1-2, 15 mg/m2/d D3-14) in 28-day cycles for 3 cycles.
  * Ph-positive B-ALL: treatment with bephytoin + TKIs, bephytoin (≥ 45 kg: 9 mcg/d D1-2, 28 mcg/d D3-14 or 28 mcg/d D1-14; < 45 kg: 5 mg/m2/d D1-2, 15 mg/m2/d D3-14) in 28-day cycles for 3 cycles.
  * Premedication with dexamethasone:
    3)For adults, premedication with dexamethasone 20 mg was administered 1 hour prior to the first dose of each cycle ofblinatumomab, prior to dose escalation (eg, Cycle 1 Day 8), and when the infusion was restarted 4 hours or more after treatment interruption.
  Pediatric patients were pre-treated with dexamethasone 5 mg/m2 up to a maximum of 20 mg prior to the first dose ofblinatumomabduring Cycle 1, prior to dose escalation (eg, Cycle 1 Day 8), and when the infusion was resumed 4 hours or more after interruption of therapy during Cycle 1
  Interventions: Drug: Blinatumomab

INTERVENTIONS:
Drug: Blinatumomab — * Ph-negative B-ALL: bephedolumab (≥ 45 kg: 9 mcg/d D1-2, 28 mcg/d D3-14 or 28 mcg/d D1-14; < 45 kg: 5 mg/m2/d D1-2, 15 mg/m2/d D3-14) in 28-day cycles for 3 cycles.
  * Ph-positive B-ALL: treatment with bephytoin + TKIs, bephytoin (≥ 45 kg: 9 mcg/d D1-2, 28 mcg/d D3-14 or 28 mcg/d D1-14; < 45 kg: 5 mg/m2/d D1-2, 15 mg/m2/d D3-14) in 28-day cycles for 3 cycles.

SUMMARY:
To explore the efficacy and safety ofblinatumomab± TKI in B-ALL patients aged ≥ 14 years with NGS-MRD relapse (sensitivity: 10-6) after auto/allo HSCT, and to observe the disease-free survival (DFS), recurrence rate and toxicity after transplantation.

DETAILED DESCRIPTION:
To explore the efficacy and safety ofblinatumomab± TKI in B-ALL patients aged ≥ 14 years with NGS-MRD relapse (sensitivity: 10-6) after auto/allo HSCT, and to observe the disease-free survival (DFS), recurrence rate and toxicity after transplantation.

Primary endpoint: disease-free survival (DFS), recurrence rate Secondary endpoints: NGS-MRD response rate, overall survival (OS), incidence of acute and chronic GVHD, and summary and evaluation of physical examination, vital signs, adverse events, concomitant treatments, and laboratory abnormalities.

* Ph-negative B-ALL: bephedolumab (≥ 45 kg: 9 mcg/d D1-2, 28 mcg/d D3-14 or 28 mcg/d D1-14; < 45 kg: 5 mg/m2/d D1-2, 15 mg/m2/d D3-14) in 28-day cycles for 3 cycles.
* Ph-positive B-ALL: treatment with bephytoin + TKIs, bephytoin (≥ 45 kg: 9 mcg/d D1-2, 28 mcg/d D3-14 or 28 mcg/d D1-14; < 45 kg: 5 mg/m2/d D1-2, 15 mg/m2/d D3-14) in 28-day cycles for 3 cycles.
* Premedication with dexamethasone:

  3)For adults, premedication with dexamethasone 20 mg was administered 1 hour prior to the first dose of each cycle ofblinatumomab, prior to dose escalation (eg, Cycle 1 Day 8), and when the infusion was restarted 4 hours or more after treatment interruption.

  4)Pediatric patients were pre-treated with dexamethasone 5 mg/m2 up to a maximum of 20 mg prior to the first dose ofblinatumomabduring Cycle 1, prior to dose escalation (eg, Cycle 1 Day 8), and when the infusion was resumed 4 hours or more after interruption of therapy during Cycle 1.

ELIGIBILITY:
Inclusion Criteria:

* 1.CD19 + acute B-lymphoblastic leukemia (Ph- or Ph + ALL); 2.Age ≥ 14 years, male or female 3.B-ALL includes any of the following:

  1. The cytogenetic prognosis of adult acute B lymphoblastic leukemia in accordance with NCCN 2023 at initial diagnosis was divided into poor prognosis group;
  2. Patients with relapsed and refractory ALL and MRD-positive ALL before transplantation,

  <!-- -->

  1. Refractory ALL is one of the following conditions. A）Failure to achieve CR/CRi at the end of induction therapy (generally referred to as 4-week regimen or Hyper-CVAD regimen).
  2. Relapsed ALL is defined as the appearance of blasts in the peripheral blood or bone marrow (> 5%), or the development of extramedullary disease in patients who have achieved CR.
  3. A positive MRD before transplantation is one of the following conditions. A）Proportion of abnormal blasts > 0.01% by flow cytometry within 45 days prior to transplantation B）Positive molecular biology related tests before transplantation; 4.NGS-IGH Conspicuous Clonal Sequences Collected (Timepoint: At initial diagnosis or prior to transplant) 5.MRD relapse (≥ 10-6, IGH-VDJ rearrangement by NGS) and < 5% bone marrow blasts at 3 and 6 months post auto/allo HSCT 6.ECOG score of 0 or 1/≤ 2 7.Adequate organ function (ALT/AST < 5 x upper limit of normal (ULN), serum bilirubin < 3.0 x ULN, creatinine clearance > 30ml/min) 8.Negative test for human immunodeficiency virus (HIV), hepatitis B surface antigen (HbsAg), and hepatitis C virus (anti-HCV) 9.Negative pregnancy test for women of childbearing potential 10.Awareness and willingness to sign written informed consent

Exclusion Criteria:

- Subjects who met any of the following criteria were not to be enrolled in the study: 6.CNSL or other extramedullary involvement after transplantation, other malignancies 7.Relevant central nervous system pathology (eg, seizure, paresis, aphasia, cerebrovascular ischemia/hemorrhage, severe brain injury, dementia, Parkinson's disease, cerebellar disease, organic brain syndrome, psychosis, or coordination or dyskinesia) 8.Co-infection active 9.Concomitant active GVHD requiring treatment 10.Product component allergy 11.Treatment with an investigational product 4 weeks prior to treatment

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
disease-free survival (DFS) | Follow-up until 3 years after transplantation
  disease-free survival (DFS)
recurrence rate | Follow-up until 3 years after transplantation
  recurrence rate

SECONDARY OUTCOMES:
NGS-MRD response rate | 3 and 6 months after transplantation and at 15 days after treatment
  Bone marrow was collected from patients at 3 and 6 months after transplantation and at 15 days after treatment with blinatumomab, and immunoglobulin rearranged IGH-VDJ sequences were monitored using high-throughput sequencing (NGS) to identify significant clonal sequences to regularly determine changes in MRD levels before and after treatment.
overall survival (OS) | Follow-up until 3 years after transplantation
  overall survival (OS)
incidence of acute and chronic GVHD | 100 days after transplantation
  The frequency and severity of acute GVHD of the intestine, skin, and liver were observed until 100 days after transplantation, and all episodes of GVHD were graded using the clinical grading criteria for acute GVHD. The changes of skin, liver function, eyes, and oral cavity of patients after 100 days after transplantation were observed to assess the incidence of localized and extensive chronic GVHD.